CLINICAL TRIAL: NCT03410875
Title: A Phase II Study of the BRAF Inhibitor, Vemurafenib, Plus Obinutuzumab in Patients With Previously Untreated Classical Hairy Cell Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-513
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hairy Cell Leukemia; Leukemia; Leukemia, Hairy Cell
Keywords: Leukemia; Hairy Cell Leukemia; BRAF; vemurafenib; obinutuzumab; Memorial Sloan Kettering Cancer Center; 17-513
MeSH Terms: conditions — Leukemia, Hairy Cell; Leukemia | interventions — Vemurafenib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Untreated Hairy Cell Leukemia (Experimental): Participants with HCL with no prior treatment for the disease
  Interventions: Drug: Vemurafenib; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Vemurafenib — Eligible patients will receive vemurafenib at a dose of 960mg orally twice daily (b.i.d.) continuously in cycles of 4 weeks (28 days) for a total of 4 cycles. In case of certain defined toxicities, dose reductions of vemurafenib by 50% (480mg b.i.d.) or interruptions of up to 15 days are permitted. If additional dose reduction is required, vemurafenib may be reduced to 240mg oral b.i.d.
Drug: Obinutuzumab — Obinutuzumab will be administered concomitantly with vemurafenib starting at cycle 2 of treatment in cycles of 4 weeks. Obinutuzumab infusions will be administered at 1000mg per day on days 1, 8 and 15 during the cycle 2 and 1000mg per day every 4 weeks during the cycle 3 and 4 of treatment.

SUMMARY:
This is a multi-center, open label, single arm, phase II trial of the oral BRAF inhibitor, vemurafenib, plus obinutuzumab in patients with previously untreated HCL. A Simon mini-max two-stage design will be employed to assess the efficacy of the combination treatment of vemurafenib and obinutuzumab. In the first stage of the protocol, 9 patients will be treated. If fewer than 6 CRs are seen among the first 9 patients, the study will be closed for lack of efficacy. If at least 7 patients respond to the treatment, then an additional 19 patients will be accrued to the second stage, for a total of 28 patients.

Eligible patients will receive vemurafenib at a dose of 960mg orally twice daily (b.i.d.) continuously in cycles of 4 weeks (28 days) for a total of 4 cycles.

Obinutuzumab will be administered concomitantly with vemurafenib starting at cycle 2 of treatment in cycles of 4 weeks. Obinutuzumab infusions will be administered at 1000mg per day on days 1, 8 and 15 during the cycle 2 and 1000mg per day every 4 weeks during the cycle 3 and 4 of treatment. After the completion of the treatment (i.e. after 4 cycles), a bone marrow aspirate and biopsy will be performed for assessment of response and evaluation of minimal residual disease (MRD). In case of certain defined toxicities, dose reductions of vemurafenib by 50% (480mg b.i.d.) or interruptions of up to 15 days are permitted. If additional dose reduction is required, vemurafenib may be reduced to 240mg oral b.i.d.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >/= 18 years of age
* Histologically confirmed classical HCL by the enrolling institution
* Has not received any prior therapy for the disease
* Patients who meet the standard treatment initiation criteria, as defined by ANC </=1.0, Hgb </=10.0 or PLT </=100K
* ECOG performance status of 0-2
* Acceptable pre-study organ function during screening as defined as:

  * Total bilirubin </= 1.5 times the upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) </=2.5x ULN
  * Serum creatinine </=1.5x ULN
* Electrocardiogram (ECG) without evidence of clinically significant ventricular arrhythmias or ischemia as determined by the investigator and a rate-corrected QT interval (QT Bazett's formula) of <480 msec
* For women of childbearing potential, agreement to the use of two acceptable methods of contraception, including one barrier method, during the study and for 6 months after discontinuation of vemurafenib
* For men with female partners of childbearing potential, agreement to use a latex condom and to advise their female partner to use an additional method of contraception during the study and for 6 months after discontinuation of vemurafenib
* Negative serum pregnancy test with 7 days of commencement of treatment in women of childbearing potential

Exclusion Criteria:

* Have had previous treatment for HCL, including purine analogs, rituximab, and other investigational agents. Previous treatment with transfusions and other supportive care such as G-CSF and erythropoietin are allowed.
* Known hypersensitivity to any of the study drugs
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
* Patients with uncorrectable electrolyte abnormalities with potassium (K) >ULN (upper limit of normal).
* Patients with any active and uncontrolled infections (such as bacterial, fungal, and new or reactivated viral infections)
* Presence of positive test results for hepatitis B virus (HBV), hepatitis B surface antigen (HBsAg) or hepatitis C (HCV) antibody.

  * Patients who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation.
  * Patients with occult or prior HBV infection (defined as positive total hepatitis B core antibody [HBcAb] and negative HBsAg) may be included if HBV DNA is undetectable. These patients must be willing to undergo monthly DNA testing.
* Known infection with HIV or human T-cell leukemia virus 1 (HTLV-1)
* Invasive malignancy that require active systemic chemotherapy or biologics that may cause significant drug-drug interaction with either vemurafenib or obinutuzumab
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Patients with HCL variant (as defined by absence of expression of CD25)
* Pregnant or lactating, or intending to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of vemurafenib in combination with obinutuzumab | 16 weeks
  Efficacy as assessed by complete response (CR) rates of participants

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Yale University, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park JH, Devlin S, Durham BH, Winer ES, Huntington S, von Keudell G, Vemuri S, Shukla M, Falco V, Cuello B, Gore S, Stone R, Abdel-Wahab O, Tallman MS. Vemurafenib and Obinutuzumab as Frontline Therapy for Hairy Cell Leukemia. NEJM Evid. 2023 Oct;2(10):EVIDoa2300074. doi: 10.1056/EVIDoa2300074. Epub 2023 Sep 21. PMID 38320179
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org